CLINICAL TRIAL: NCT07137260
Title: Digital Assessment of Real-World Walking Activity in Pulmonary Hypertension: A Prospective Multicenter Trial
Status: Recruiting | Type: Observational
Sponsor: Simon Jäger (Other)
Collaborators: Klinikum Nürnberg (Other); LMU Klinikum (Other); SLK Kliniken Heilbronn GmbH (Other); Robert Bosch Medical Center (Other)
Responsible Party: Sponsor-Investigator, Simon Jäger, Head: Institute of Clinical Pharmacology, Paracelsus Medical University
Organization: Paracelsus Medical University (Other)
Other Study IDs: CPN_PMU001
Record Dates: First submitted 2025-07-09; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Pulmonary Hypertension; Precapillary Pulmonary Hypertension; Right Heart Catheterisation; Digital Mobility Outcomes
Keywords: Digital mobility assessment; Right heart catheterization; Mobility assessment; Digital mobility outcome; Pulmonary hypertension; Pulmonary arterial hypertension; Sensor; Axivity sensor; Precapillary pulmonary hypertension; Walking assessment; Walking test; Physical activity
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Arterial Hypertension; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients newly diagnosed with precapillary pulmonary hypertension: Diagnosis of precapillary pulmonary hypertension confirmed by right heart catheterization (as described under inclusion criteria) with follow-up visits planned by the treating clinician in the next 3-12 months.
  Interventions: Device: Accelerometer (measurement of walking activity)

INTERVENTIONS:
Device: Accelerometer (measurement of walking activity) — Wearing an accelerometer (size 23x32,5x8,9 mm, weight 11g) on the lower back consistently for one week at a time to measure walking activity. The sensor is fixed with waterproof plasters. No feedback is given to the participant while wearing the sensor and no data can be read directly from the sensor.

SUMMARY:
The goal of this observational study is to validate digital mobility outcomes for monitoring the treatment and disease progression in adult patients with pulmonary hypertension. The main question it aims to answer is:

-Do digital mobility outcomes (measured digital endpoints characterizing walking behavior) correlate with measures of precapillary pulmonary pressure as assessed by right heart catheterization?

Participants will be asked to wear a small sensor on the lower back for one week at a time for a total of 3 times: at diagnosis and follow-up visits at 3-6 months and again at 6-12 months. Follow-up visits are scheduled by the treating clinician. At the end of the study participants can choose to receive feedback on the sensor measurements.

ELIGIBILITY:
Inclusion Criteria:

* Pulmonary hypertension confirmed by right heart catheterization
* Presence of precapillary pulmonary hypertension at time of recruitment, defined as mean pulmonary arterial pressure (MAP) ≥ 20 mmHg, pulmonary arterial wedge pressure (PAWP) ≤ 15 mmHg and pulmonary vascular resistance (PVR) > 2 Wood units (160 dyn·s·cm-5)
* After the right heart catheterization another follow-up visit is required in 3, 6, or 12 months
* Independent walking without assistance and a 6-min walking distance > 100m
* WHO Functional Class I-III
* Ability to provide informed consent and to participate in the study procedures
* Willingness to wear the Axivity AX6 Sensor for 7 days

Exclusion Criteria:

* Hospitalization for a pulmonological disease within the 30 days prior to study recruitment
* Neurological or orthopedic disease which limits walking ability
* Acute pain which limits walking ability
* Poor vision, which limits walking ability
* Terminal illness with life expectancy < 1 year
* Ongoing treatment for malignancy
* Acute psychosis or other severe psychiatric illness
* Substance dependence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with precapillary pulmonary hypertension and receiving treatment at participating study centres.
Sampling Method: Non-Probability Sample
Enrollment: 77 (Estimated)
Dates: Start 2024-04-19 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Correlation of digital mobility assessments with measured pulmonary arterial pressures | Baseline assessment at first diagnosis, follow-up assessments after 3-6 months and again after 6-12 months (follow-up time frames are determined by the treating clinician).
  Correlation of the digital mobility and walking parameters measured by the Axivity AX6 sensor with the precapillary pulmonary artery pressure during right heart catheterization. As the digital mobility parameters for pulmonary hypertension are still largely unknown, the primary variable will be the average walking speed for walking episodes of > 30 seconds and compared with the measured pulmonary vascular resistance. The sensor is worn for 1 week at a time for a total of three sets of measurements (determined by scheduled clinical follow-up visits). The goal is to determine the feasibility of digital parameters for risk stratification and measuring disease activity and response to treatment.

SECONDARY OUTCOMES:
Description of the general daily walking behaviour of patients with precapillary pulmonary hypertension: amount of walking episodes | Measured at diagnosis (baseline visit) and two follow-up visits (between 3-6 months and again after 6-12 months, as determined by the treating clinician).
  Amount of walking episodes as measured by the AX6 Axivity Sensor. The sensor is worn on the lower back for 1 week at a time at diagnosis and two follow-up visits.
Description of the general daily walking behaviour of patients with precapillary pulmonary hypertension: duration of walking episodes | Measured at diagnosis (baseline visit) and two follow-up visits (between 3-6 months and again after 6-12 months, as determined by the treating clinician).
  Duration of walking episodes in seconds, hours and minutes as measured by the AX6 Axivity Sensor. The sensor is worn on the lower back for 1 week at a time at diagnosis and two follow-up visits.
Description of the general daily walking behaviour of patients with precapillary pulmonary hypertension: amount of steps | Measured at diagnosis (baseline visit) and two follow-up visits (between 3-6 months and again after 6-12 months, as determined by the treating clinician).
  Amount of daily steps as measured by the AX6 Axivity Sensor. The sensor is worn on the lower back for 1 week at a time at diagnosis and two follow-up visits.
Correlation between validated digital mobility outcomes and important prognostic markers of cardiac function | Measured at diagnosis (baseline visit) and two follow-up visits (between 3-6 months and again after 6-12 months, as determined by the treating clinician).
  Correlation of validated digital mobility outcomes with prognostic markers of cardiac function:
  * Right heart catheterization: middle pulmonary arterial pressure, right atrial pressure, cardiac index, mixed venous saturation
  * Echocardiography: right atrial size, systolic pulmonary artery pressure (SPAP), Tricuspid annular plane systolic excursion (TAPSE)
  * NT-proBNP
Correlation between digital mobility outcomes and disease progression | Measured at diagnosis (baseline visit) and two follow-up visits (between 3-6 months and again after 6-12 months, as determined by the treating clinician).
  Correlation between validated digital mobility outcomes and clinical progression of pulmonary hypertension. Disease progression is measured by mortality, hospital admission secondary to pulmonary hypertension, and changes in any of the following: WHO functional class, REVEAL score (Registry Risk Score for Pulmonary Arterial Hypertension), COMPERA score (Comparative, Prospective Registry of Newly Initiated Therapies for Pulmonary Hypertension), dyspnea (mMMRC), emPHasis-10 score, 6-minute walking test.
Investigation of potential confounders | From enrollment to end of study after the last follow-up visit at 6-12 months.
  Investigation of potential confounders such as functional capacity (6-minute walking test, WHO functional class), sex, age, mono-, dual-, or tripple therapy for pulmonary hypertension.

CONTACTS AND LOCATIONS:
Locations (4):
- Germany (4):
  - Robert Bosch Hospital, Stuttgart, Baden-Wurttemberg
  - Internal Medicine Clinic V, Ludwig-Maximilians-University Clinic, Munich, Bavaria
  - Klinikum Nuremberg, Nuremberg, Bavaria
  - SLK-Kliniken Heilbronn GmbH - Fachklinik Löwenstein, Löwenstein

IPD SHARING:
Plan to Share IPD: No